CLINICAL TRIAL: NCT02052102
Title: A Cohort Study Assessing Cardiac Function With MRI in Left-Sided Breast Cancer Patients Treated With Deep Inspiration Breath Hold (DIBH) Technique to Improve Cardiac Sparing During Adjuvant Radiotherapy
Brief Title: Study to See Whether Breath-Hold Techniques During RT Are Effective in Helping to Improve Sparing of the Heart
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Breast-26159
Record Dates: First submitted 2014-01-24; First posted 2014-01-31 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer; Adverse Effect of Radiation Therapy
Keywords: Deep inspiration breath hold; radiation therapy; Cardiac toxicity; Left-sided breast cancer
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries; Cardiotoxicity; Unilateral Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No prior therapy, DIBH irradiation (Active Comparator): Cohort 1 - No prior anthracycline-based chemotherapy or herceptin, deep inspiration breath hold breast radiation therapy
  Interventions: Radiation: Radiation therapy
- No prior therapy, FB technique (Active Comparator): Cohort II - no prior Anthracycline based chemotherapy or Herceptin and (ii) to receive FB RT (not able to hold breath for at least 20 seconds or does not have a minimum of 1.0 cm of heart on at least 3 slices (3mm slices) on the FB scan)
  Interventions: Radiation: Radiation therapy
- Prior therapy, DIBH irradiation (Active Comparator): Cohort III - Prior Anthracycline-based chemotherapy or Herceptin, and (ii) eligible to receive DIBH RT. (Patient has a minimum of 1.0 cm of heart on at least 3 slices (3mm slices) on the FB scan)
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Radiation: Radiation therapy

SUMMARY:
The study hopes to determine whether patients with left-sided breast cancer are at an increased risk of cardiac changes due to radiation to the breast +/- Anthracycline-based chemotherapy +/- Herceptin and whether a deep inspiration breath hold (DIBH) technique during radiotherapy treatments would further reduce dosimetric dose to the heart as compared to the conventional free breathing (FB) technique thus reducing cardiac toxicity as measured by cardiac MRI using left ventricular end-diastolic volume (LVEDV) as a metric. Bio fluid samples will also be collected to investigate specific biomarkers of breast cancer: BNP, PIIINP and CITP

DETAILED DESCRIPTION:
Patients with left-sided breast cancer who receive adjuvant breast or chest wall radiation have increased risk of treatment related cardiovascular morbidity. The risk of cardiac morbidity and mortality is increased when a patient receives radiation following adjuvant chemotherapy and Herceptin. The dose-volume histogram (DVH) parameters associated with increased cardiac toxicity include volume of heart irradiated, total radiation dose received by the left ventricle (LV), V25 and mean cardiac dose. Even though modern RT treatments like 3DCRT and IMRT can reduce the mean dose to the heart, the maximum dose to the left side of the heart/LV may not be reduced if the target is close to the heart. The hypothesis is that DIBH RT can safely and effectively reduce the heart dose, especially the dose to the LV, that could lead to reduction in the incidence of radiation induced cardiovascular morbidity and mortality.

Radiotherapy has detrimental effects on cardiac function due to remodeling of the cardiac tissue that receive radiation. We believe that the radiation related acute effects on heart tissue can be detected with cardiac functional MRI. The study will quantify the acute RT related effects. To our knowledge, cardiac MRI has not been explored as a non invasive technique to quantify RT +/- chemotherapy related effects.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with pathologically confirmed left sided breast cancer eligible for adjuvant breast/chest wall plus or minus regional nodal radiotherapy
* Women patients with age group between 18 and 70 years old
* Karnofsky performance score ≥ 70
* Ability to hold breath for at least 20 sec (for DIBH cohorts only)
* Life expectancy >10 years

Exclusion Criteria:

* For patients with prior Anthracycline based chemotherapy or Herceptin, if there is < 1.0 cm of heart on at least 3 slices ( 3 mm slices) on the FB scan, the patient will be considered a screen failure.
* Previously irradiated or recurrent breast/chest wall tumours or previous malignancy other than non-melanoma skin cancer unless disease free for a minimum of 5 years prior to study entry
* Patients that require a shell for breast immobilization
* Patients requiring a boost
* Stage IV disease

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-02 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Radiation related acute and long term functional changes in patients treated with deep-inspiration breath hold compared to free-breathing technique | 12 months
  Using MRI-based cardiac functional imaging to measure radiation-related acute and long term cardiac functional changes in patients treated with deep-inspiration breath-hold (DIBH) compared to free breathing (FB) treatment

SECONDARY OUTCOMES:
Radiation dosimetric comparison | 12 months
  Radiation dosimetry is the accurate calculation and measurement of radiation doses received by tissue resulting from the exposure to radiation. A radiation dosimetric comparison will be performed between the deep inspiration breath hold (DIBH) technique treatment plan and the free breathing (FB) technique treatment plan to explore sparing of cardiac sub-structures from radiation, if any

CONTACTS AND LOCATIONS:
Overall Officials: Kurian Joseph, MB, FFRRCSI, FRCR, FRCPC, Principal Investigator — Cross Cancer Institute
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No